CLINICAL TRIAL: NCT03999567
Title: A Validation Study of a Mobile Phone Digit Symbol Substitution Test Application for Cognition in Adults With Major Depressive Disorder
Brief Title: Validation Study: Mobile DSST on Cognition in Adults With MDD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brain and Cognition Discovery Foundation (Other)
Collaborators: Takeda (Industry); Cognition Kit (Unknown); Ctrl Group, Ltd (Unknown)
Responsible Party: Principal Investigator, Dr. Roger S. McIntyre, Chairman and Executive Director, Brain and Cognition Discovery Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00037042
Record Dates: First submitted 2019-06-20; First posted 2019-06-26 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Major Depressive Episode
MeSH Terms: interventions — penclomedine

STUDY DESIGN:
Intervention Model Description: Thirty adults (18-65) with DSM-5 MDD will be enrolled at the BCDF Toronto, Ontario. All subjects will have their diagnosis confirmed by Mini International Neuropsychiatric Interview Version 6.0.
  At baseline, data will be collected from all participants and will include demographics, comorbidities, medication history and concurrent medications. All subjects will be assessed symptomatically with the Montgomery and Asberg Depression Rating Scale (MADRS) as well as the Hamilton Anxiety Rating Scale (HAM-A), Snaith Hamilton Pleasure Scale (SHAPS) for anhedonia, as well as the paper and pencil version of the DSST at baseline and end of study (Day 7).
  The DSST has been normed on the sex, age and gender. These norms will be used as reference. All subjects will complete the pencil and paper version of the DSST and complete the mobile app-based version of the DSST.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pen and Paper vs. Mobile Digit Symbol Substitution Test (Experimental): This validation study will assess the convergent validity of the mobile DSST application with the pencil version of the DSST. Correlations between performance on app-based version of the DSST and paper-based version of DSST will be measured.
  Interventions: Other: Pen and Paper Digit Symbol Substitution Test (DSST); Other: Electronic Digit Symbol Substitution Test (DSST)- (a.k.a. Codebreaker)

INTERVENTIONS:
Other: Pen and Paper Digit Symbol Substitution Test (DSST) — The DSST is a paper-and-pencil cognitive test presented on a single sheet of paper that requires a subject to match symbols to numbers according to a key located on the top of the page. The subject copies the symbol into spaces below a row of numbers. The number of correct symbols within the allowed time, usually 90 to 120 seconds, constitutes the score.
Other: Electronic Digit Symbol Substitution Test (DSST)- (a.k.a. Codebreaker) — Code breaker is the mobile/electronic version of the pen and paper DSST which is capable of identifying deficits in the domains of executive function, processing speed and attention/concentration, and takes 2 minutes to complete. Six symbols are numbered consecutively. Users are presented with a series of numbers that they must then match with the correct corresponding symbol as quickly as possible. Users are scored on speed and accuracy.

SUMMARY:
Objectives The primary objective of this study is to determine the convergent validity of the mobile DSST application with the pencil and paper version of the DSST.

Design and Outcomes This study will be performed by the Brain and Cognition Discovery Foundation (BCDF). The BCDF is an organization based in Toronto, Ontario, Canada led by Dr. Roger S. McIntyre. Membership of the BCDF has developed and validated rating scales and metrics for adults with mood disorders for over 10 years. A member of the BCDF provides diagnoses and treatment for adults (age 18-65) with mood disorders and provides clinical care to the largest catchment area in Canada. The BCDF conducts clinical research according to the International Conference on Harmonization, Declaration of Helsinki, and Good Clinical Practice (GCP) guidelines. The study will be approved by the community Research Ethics Board.

Thirty adults (18-65) with DSM-5 MDD will be enrolled at the BCDF Toronto, Ontario. All subjects will have their diagnosis ascertained clinically and confirmed by Mini International Neuropsychiatric Interview Version 5.0 (M.I.N.I.).

At baseline, data will be collected from all participants and will include demographics, comorbidities, medication history and concurrent medications. All subjects will be assessed symptomatically with the Montgomery and Asberg Depression Rating Scale (MADRS) as well as the Hamilton Anxiety Rating Scale (HAM-A), Snaith Hamilton Pleasure Scale (SHAPS) for anhedonia, as well as the paper and pencil version of the DSST at baseline and end of study (Day 7).

The DSST has been normed on the sex, age and gender. These norms will be used as reference. All subjects will complete the pencil and paper version of the DSST and complete the mobile app-based version of the DSST.

Sample Size and Population This is a small validation study of 30 subjects. Subjects diagnosed with major depressive disorder will be eligible for participation in this study.

DETAILED DESCRIPTION:
Primary Objective The primary objective of this study is to determine the convergent validity of the mobile DSST application with the pencil version of the DSST.

Secondary Objectives To determine whether a correlation exists between the digitalized DSST performance and depression symptoms severity.

To determine patient satisfaction with the digitalized version of the DSST as measured by a satisfaction Likert scale.

Background Health-related information and communication technology solutions that utilize mobile phones, known as mobile health applications (apps), have the potential to expand health interventions beyond face-to-face contacts of traditional healthcare. For the healthcare provider, mobile apps can offer low cost and easily scalable interventions to monitor and improve services to patient populations that are difficult to retain in treatment, potentially leading to more sensitive measurement of cognition, mood and may promote better health. Uptake of health-related mobile apps has increased in recent years as technology barriers such as access, knowledge, and product usability have improved, reducing obstacles for 'digitally excluded' subpopulations (e.g., poor, rural, and older). Consensus exists that the availability of a mobile phone application-based cognitive measure would be more user friendly, aligned with busy office practice and would be more likely to be adopted by end users. Patients with depression and their treating provider may benefit from the use of a mobile health app to assist in disease self-management. This validation study will assess the convergent validity of the mobile DSST application with the pencil version of the DSST. Correlations between performance on app-based version of the DSST and paper-based version of DSST will be measured.

Study Rationale MDD is a serious public health concern worldwide with ample documentation demonstrating that MDD is one of the leading contributors to the global burden of disease and is currently the leading cause of disability worldwide. Moreover, the economic burden of MDD is estimated to total $210.5 billion with approximately 50% of the cost being attributable to impairment in role function (e.g., workplace performance: presenteeism, absenteeism, and short-/long-term disability). Accumulating evidence suggests that the treatment and resolution of mood symptoms among individuals with MDD is insufficient in facilitating full functional recovery among individuals affected by MDD wherein a highly reproduced observation is that impairments in cognitive function remain persistent, pervasive, and progressive during the "remitted" state. The foregoing portrait of MDD as a multidimensional syndrome associated with cognitive impairment and differential functional implications, provides the impetus for evaluating the disparate domains commonly affected in this clinical population using valid and reliable measures/assessments capable of providing actionable information in the treatment and management of patients.

Hitherto, clinical awareness surrounding the pertinence of cognitive impairment in MDD and its impact on functional recovery has been limited with no "gold standard tool(s)" to detect cognitive impairments in adults with MDD. Moreover, although several screening/measurement instruments are currently available that have demonstrated sensitivity to cognitive impairments in select cognitive domains, only one tool, to the authors' knowledge, has been developed primarily to evaluate the four principal cognitive domains affected in adults (18-65) with MDD (i.e., executive function, learning and memory, processing speed, as well as attention/concentration) using a composite score.

Available evidence, and evidence-based guidelines for MDD now recommend systematic assessment and measurement of cognitive dysfunction in adults with MDD. A barrier to implementation of the foregoing recommendation is the availability of a user-friendly point of care patient administered potentially interoperable engaging measure of cognitive function with in MDD.

Although many screening instruments and neurocognitive batteries are available to assess cognition, most are not routinely available in clinical ecosystems and/or are costly, require professional interpretation and/or too cumbersome for busy office practice.

STUDY DESIGN This study will be performed by the BCDF. The BCDF is an organization based in Toronto, Ontario, Canada led by Dr. Roger S. McIntyre. Membership of the BCDF has developed and validated rating scales and metrics for adults with mood disorders for over 10 years. A member of the BCDF provides diagnoses and treatment for adults (age 18-65) with mood disorders and provides clinical care to the largest catchment area in Canada. The BCDF conducts clinical research according to the International Conference on Harmonization, Declaration of Helsinki, and GCP guidelines. The study will be approved by the community Research Ethics Board.

Thirty adults (18-65) with DSM-5 MDD will be enrolled at the BCDF Toronto, Ontario. All subjects will have their diagnosis ascertained clinically and confirmed by MINI.

Study Enrollment Procedures Upon identifying a subject who meets the criteria for study participation, the physician providing care for that subject, or the coordinator acting on behalf of the physician with the physician's consent, will explain the study, answer any questions about the study and obtain informed consent.

Study participants will be compensated a total of $400 for participation in this 1-week study, $0.00 at the time of completion of baseline assessments, and $400 at the time of completion of the end of study assessments.

STUDY INTERVENTIONS The interventions in this study include a mobile health app, completion of pencil and paper DSST. Subjects will then complete the app-based version of the DSST.

Description of Study Evaluations Consenting Procedure Eligible subjects will be recruited from the BCDF. All eligible subjects will engage in a thorough consenting process as it relates to the aims, objectives and hypotheses of the study. The voluntariness of all eligible subjects will be emphasized, and participation/ non-participation will have no impact on care recommendations. Upon completion of the consenting process, all eligible subjects will be asked to sign a consent form at the BCDF. Patients who are eligible will be explained the details of the study by the treating physician and will be provided with the opportunity to ask any questions before consent is obtained. A research study coordinator will explain the study and obtain and document consent using a Medical Ethics Board (MEB) approved consent form.

Screening Screening of subjects for eligibility will be performed by research study staff and treating physicians either prior to the subject's visit or at the time of the visit. Subjects with MDD, as confirmed using M.I.N.I Version 5.0, who meet all the selection criteria are eligible for participation.

Study Visits The study will consist of two visits, baseline and final visit. The paper DSST and the mobile app DSST will be completed at each of these visits. MADRS, HAM-A and SHAPS assessments will also be completed at baseline and final visit.

Completion/Final Evaluation/Early Termination Subjects will complete a final visit. All eligible subjects will be informed that the ongoing provision of care will not be guaranteed. Necessary steps will be put in place to assure that subjects are made aware of mental health resources for ongoing care in emergency situations.

ELIGIBILITY:
Inclusion Criteria:

* The participant is able and willing to provide informed consent.
* The participant is male or female 18-65 years of age and owns a smart phone.
* The participant has received a current diagnosis of a major depressive episode (MDE) as part of MDD as per DSM-5 criteria.
* The participant's current MDE is confirmed by the M.I.N.I.
* The participant is an outpatient of a psychiatric setting.
* The participant has a MADRS score ≥ 20 at screening and baseline.
* At least one prior MDE formally diagnosed by a healthcare provider or validated by previous treatment (e.g., guideline-informed pharmacotherapy and/or manual-based psychotherapy).

Exclusion Criteria:

* Current alcohol and/or substance use disorder as confirmed by the M.I.N.I.
* Presence of comorbid psychiatric disorder other than MDD that is a focus of clinical concern as confirmed by the M.I.N.I.
* Medications approved and/or employed off-label for cognitive dysfunction (e.g., psychostimulants).
* Any medication for a general medical disorder that, in the opinion of the investigator, may affect cognitive function.
* Use of benzodiazepines within 12 hours of cognitive assessments.
* Consumption of alcohol within 8 hours of cognitive assessments.
* Inconsistent use or abuse of marijuana.
* Physical, cognitive, or language impairments sufficient to adversely affect data derived from cognitive assessments.
* Diagnosed reading disability or dyslexia.
* Clinically significant learning disorder by history.
* Electroconvulsive therapy (ECT) in the last 6 months.
* History of moderate or severe head trauma (e.g., loss of consciousness for >1 hour), other neurological disorders, or unstable systemic medical diseases that in the opinion of the investigator are likely to affect the central nervous system.
* Pregnant and/or breastfeeding.
* Received investigational agents as part of a separate study within 30 days of the screening visit.
* Actively suicidal/presence of suicidal ideation or evaluated as being a suicide risk (as per clinical judgment using the Columbia-Suicide Severity Rating Scale).
* Currently receiving treatment with Monoamine Oxidase Inhibitors anti-depressants, antibiotics such as linezolid, or intravenous methylene blue.
* Previous hypersensitivity reaction to vortioxetine or any components of the formulation.
* Clinical worsening symptoms of depression and suicide risk based on investigator judgement.
* History of or current diagnosis of Serotonin syndrome.
* History of or current Abnormal bleeding.
* Previous history or current symptoms of mania/hypomania.
* Angle closure glaucoma.
* Hyponatremia.
* Moderate hepatic impairment.
* History of seizures and epilepsy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-08-25 (Actual); Primary Completion 2020-02-04 (Actual); Study Completion 2020-02-04 (Actual)

PRIMARY OUTCOMES:
Validation of the mobile DSST application | 1 week
  The primary objective of this study is to determine the convergent validity of the mobile DSST application with the pencil version of the DSST. Correlation between performance on the digitalized DSST and the pencil and paper version will be conducted. In light of the small sample size and this being a feasibility pilot study, we will be looking at descriptive statistics of demographics, depression severity and cognition performance. An interim analysis will be completed after the first 15 subjects complete the study.

SECONDARY OUTCOMES:
Montgomery and Asberg Depression Rating Scale (MADRS) | 1 week
  Scale that assesses depressive symptoms. The scale has 10 items and is based on the patient's subjective report of his/her clinical condition over the previous 7 days. Additional information is based upon clinical observations made during the course of the clinical interview. Each item assesses a severity rating. All items that are graded on a 0 to 6 scale. The overall MADRS score ranges from 0-60. Higher scores are indicative of more severe depression.Usual cutoff points are: 0 to 6 - normal/symptom absent; 7 to 19 - mild depression; 20 to 34 - moderate depression; >34 - severe depression.
Hamilton Anxiety Rating Scale (HAM-A) | 1 week
  The HAM-A is a rating scale that measures the severity of anxiety symptoms.The scale consists of 14 items, each defined by a series of symptoms, and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety).
Snaith Hamilton Pleasure Scale (SHAPS ) | 1 week
  The SHAPS is a 14-item scale that measures anhedonia, the inability to experience pleasure. The items cover the domains of: social interaction, food and drink, sensory experience, and interest/pastimes. A score of 2 or less constitutes a "normal" score, while an "abnormal" score is defined as 3 or more. Each item has four possible responses: strongly disagree, disagree, agree, or strongly agree. Either of the "disagree" responses score one point, and either of the "agree" responses score 0 points. Thus, the final score ranges from 0 to 14 and higher scores are indicative of greater anhedonia.

CONTACTS AND LOCATIONS:
Overall Officials: Roger McIntyre, MD, Principal Investigator — Brain and Cognition Discovery Foundation
Locations (1):
- Canadian Rapid Treatment Centre of Excellence, Mississauga, Ontario, Canada

REFERENCES:
- [Derived] McIntyre RS, Lipsitz O, Rodrigues NB, Subramaniapillai M, Nasri F, Lee Y, Fehnert B, King J, Chrones L, Kratiuk K, Uddin S, Rosenblat JD, Mansur RB, McCue M. An App-Based Digit Symbol Substitution Test for Assessment of Cognitive Deficits in Adults With Major Depressive Disorder: Evaluation Study. JMIR Ment Health. 2022 Oct 27;9(10):e33871. doi: 10.2196/33871. PMID 36301615